CLINICAL TRIAL: NCT01536236
Title: A Randomized, Comparison Study of the Safety and Efficacy of Spinal Cord Stimulation Versus Standard of Care Medical Management in the Treatment of Diabetic Polyneuropathy
Brief Title: Spinal Cord Stimulation for Diabetic Polyneuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRD_505
Record Dates: First submitted 2011-10-17; First posted 2012-02-20 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Polyneuropathy
Keywords: Diabetes; Polyneuropathy; Spinal cord stimulation
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Polyneuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subthreshold programming (Active Comparator): During one of the first 2 weeks of the trial the subject will be randomized to a subthreshold stimulation arm. They will be blinded and receiving therapy, but will it will be delivered at a level (subthreshold) that they will not feel the stimulation.
  Interventions: Device: ANS Eon™ Implantable Pulse Generator (Permanent Implant)
- Placebo or Stimulation off arm (Placebo Comparator): During one of the first two weeks of the study, the patient will be randomized to a no stimulation arm. They will be blinded and will not be receiving therapy.
  Interventions: Device: ANS Eon™ Implantable Pulse Generator (Permanent Implant); Device: Placebo
- Optimal stimulation programming (Active Comparator): During the third week of the trial period, all subjects will receive optimal stimulation.
  Interventions: Device: ANS Eon™ Implantable Pulse Generator (Permanent Implant)

INTERVENTIONS:
Device: ANS Eon™ Implantable Pulse Generator (Permanent Implant) — Appropriate programming based on subject's preference of programs.
Device: Placebo — Placebo
  Arms: Placebo or Stimulation off arm

SUMMARY:
To obtain preliminary estimates of the safety and efficacy of the ANS Eon™ Implantable Pulse Generator with ANS leads in the treatment of subjects with diabetic polyneuropathy.

DETAILED DESCRIPTION:
There is a medication arm and a stimulation arm. Patients will randomized to one or the other. If patients are randomized to the medication arm, after 6 months they have the option of going into the stimulation arm. There is a 3 week trial which includes a crossover period from "no stimulation" to subthreshold stimulation. The 3rd week patients will receive "optimal" stimulation. If they qualify, they will be implanted with the permanent device.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years of age or older
2. The subject has signed and received a copy of an informed consent form after the nature of the study has been fully explained.
3. The subject has a clinical diagnosis of diabetes mellitus
4. The subject has an A1C less than or equal to 10% within the last 3 months.
5. The subject has been on a stable diabetic therapy for at least 3 months without hospitalizations for control of diabetes.
6. The subject has a documented clinical diagnosis of painful diabetic distal symmetric sensory/motor polyneuropathy using the LANSS (Leeds assessment of neuropathic symptoms and signs) pain scale score of 12 or greater and the TNS (total neuropathy score) score of 20 or greater.
7. The subject has bilateral, moderate to severe pain from diabetic polyneuropathy for the previous 3 months.
8. The subject has a VAS of > 4 at Baseline, on a stable analgesic regimen consisting of any one or combination of the following agents: anticonvulsants, antidepressants, and opioids for 1 month.
9. The subject has been shown to be refractory to conservative therapy by failing a minimum of 3 conservative treatments at least one of which is a medication specifically for diabetic polyneuropathy of adequate dose and duration
10. Female subject has a negative pregnancy test.

Exclusion Criteria:

1. Subject is unwilling or unable, in the opinion of the investigator, to comply with study instructions.
2. Subject has other severe pain that could confound the assessment of pain due to diabetic polyneuropathy.
3. Subject has a neuropathy that the investigator considers is not due to diabetes (e.g., significant vasculitis, collagen vascular disorder, medications known to cause neuropathies, history of familial neuropathy, drug or alcohol abuse, hepatitis, HIV, infection or pernicious anemia)
4. Subject has had any amputation.
5. Subject has a diagnosis within the past 1 year of major psychiatric disturbance. Exclusionary psychiatric diagnoses include the following Axis I disorders (DSM-IVR criteria): major depression, bipolar disorder, schizophrenia or other psychotic disorder or somatoform disorders. The Axis II disorder of borderline personality is also excluded.
6. Subject has co-existent, major systemic disease(s) that would interfere with interpretation of study results (e.g. malignancy, poorly controlled diabetes, ischemic cardiac disease, profound autonomic dysfunction or any other disease in the opinion of the investigator.)
7. Subject who has an abnormal PT, PTT, bleeding time or platelet count that might interfere with therapy.
8. Subject is currently participating in or has, within the past 30 days, participated in a study of another investigational drug or device.
9. Subject has a history of substance abuse within the past 2 years.
10. Subject has a demand-type pacemaker or implanted cardiac defibrillator.
11. Subject who require diathermy or MRIs.
12. Subject with any metallic implants that might interfere with this therapy in the opinion of the investigator;
13. Subject who has an implanted medication pump or implanted neurostimulation device.
14. Subject who currently has an active infection.
15. Subject who currently has foot ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 24 months
  The VAS is a 100mm line that indicates severity of pain progression

SECONDARY OUTCOMES:
Device related and serious adverse events | 24 months +/- 6 months depending on study arm randomization
  All adverse events that are classified as device related and/or serious will be assessed.
Neuropathy Impairment in the Lower Limbs (NIS-LL) | 24 months
  Neuropathy Impairment Score in the Lower Limbs (NIS-LL):
  The NIS-LL is a quantitative neurological examination that evaluates changes in motor, sensory and reflex activity in the lower limbs. The test has 14 items: 8 to evaluate muscle strength (64 possible points), 2 items to evaluate reflex activity (8 possible points), and 4 items to evaluate sensory activity (16 possible points). All items are tested bilaterally and the maximum score is 88 points.
Nerve conduction studies and Electromyogram (EMG) | 24 months
  Electromyography (EMG) is a technique for evaluating and recording the electrical activity of muscles. This test will be performed according to standard practice.
Inflammatory mediators (IL-6, IL-1β, and CRP) | 24 months
  A complete blood count (CBC), comprehensive metabolic panel (CMP) and PT, (Prothrombin Time), PTT (Partial Thromboplastin Time) will be performed as well as assessment of hemoglobin A1c (HbA1c), interleukin-6 (IL-6), interleukin-1 beta (IL-1β), and C-reactive protein (CRP) levels. HbA1c is used to evaluate the amount of glycosylated hemoglobin in the blood which is indicative of blood glucose levels. IL-6 and IL-1β, and CRP are indicators of an inflammatory response and are consistently associated with diabetic polyneuropathy.
Vascular Doppler | 24 months
  A Doppler ultrasound uses reflected sound waves to evaluate blood as it flows through the major arteries and veins of the arms, legs, and neck. This test will be performed according to standard practice.
Intra-epidermal skin biopsy | 24 months
  A skin biopsy will be performed to assess damage to nerve fibers due to DPN.
Short Form 36 (SF-36) Quality of Life Questionnaire | 24 months
  The SF-36 is a 36-item tool for measuring health related quality of life from the patient's point of view. The items on the questionnaire are scored and divided into 8 sub-scales, and each subscale is also categorized as a physical component or a mental component.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Diaz, Study Director — Abbott Medical Devices
Locations (1):
- Midwest Neurosurgery Associates, Kansas City, Missouri, United States